CLINICAL TRIAL: NCT06416878
Title: Can Brief Perioperative Epidural Electrical Stimulation Improve Recovery of Autonomic Function in Cauda Equina Syndrome
Brief Title: Brief ES for Recovery of Autonomic Function in CES
Acronym: BESCES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UoL001787
Record Dates: First submitted 2024-01-08; First posted 2024-05-16 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Cauda Equina Syndrome
Keywords: cauda equina syndrome; electrical stimulation; spinal cord stimulator; recovery of autonomic function; axonal regeneration
MeSH Terms: conditions — Cauda Equina Syndrome

STUDY DESIGN:
Intervention Model Description: Consecutive patients presenting to neurosurgical department with acute cauda equina syndrome with autonomic dysfunction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): All participants
  Interventions: Device: Brief ES at the time of decompression for cauda equina syndrome; Device: Brief ES to facilitate mcturition/removal of catheter

INTERVENTIONS:
Device: Brief ES at the time of decompression for cauda equina syndrome — In patients operated for acute cauda equina syndrome with autonomic dysfunction epidural ES will be delivered utilising SCS trial electrode. It will be delivered for 10 minutes caudal to compression site and for 60 mins cranial to compression site while the wound is closed and patient recovered.
Device: Brief ES to facilitate mcturition/removal of catheter — In patients who do not fully recover function following decompression, brief ES will be applied before second micturition attempt.

SUMMARY:
BESCES is a study that aims to explore the feasibility of intraoperative brief epidural electrical stimulation (ES) for patients undergoing routine decompression for cauda equina syndrome. In consenting patients, brief ES will be applied using a CE-marked SCS trial kit once sufficient decompression is achieved. In participants who do not recover function following decompression, brief post-op ES will be applied to see if can facilitate micturition and/or removal of the catheter.

The study will assess:

The feasibility of intervention. If brief ES can facilitate conduction in residual neurons. If brief ES can facilitate neuronal recovery

DETAILED DESCRIPTION:
Cauda equina syndrome (CES), defined as a compression of nerves controlling bowel, bladder and sexual function due to lumbar disc prolapse has a prevalence of 2 per 100,000 UK population per year. It mostly affects individuals 30-49 years of age. Emergency surgery to decompress the nerves is the mainstay of treatment. Despite adequate decompression, 17% of patients are left incontinent and 50% experience persistent bowel, bladder or sexual dysfunction needing long-term supportive symptomatic management and compromising their social cohesion and economic productivity.

Theoretically, there are two possible ways of improving these functions - improving regeneration of damaged cells and improving conduction in partially damaged/residual cells. The use of perioperative electrical stimulation (ES) has shown significant promise in facilitating recovery in peripheral nerve compression syndromes. Epidural stimulation is routinely used for treating neuropathic pain and there is anecdotal evidence of improved bladder and bowel function in patients with CES who have received epidural spinal cord stimulation for chronic pain.

The overall aim of this feasibility study is to determine if a full definitive RCT is possible. The investigators want to see if it is possible to timely and safely deliver epidural stimulation in patients presenting with bowel, bladder or sexual dysfunction due to cauda equina compression, undergoing emergency lumbar decompression, assess the potential effect size of brief post-decompression ES proximal to the level of compression in facilitating axonal regeneration to support further RCT. The investigators also want to see if brief ES can improve conduction in residual neurons.

40 patients presenting with CES shall be enrolled. At the time of decompression surgery, consenting patients shall receive ES. With standard care, patients who still have symptoms after decompression, remain symptomatic at 1 year. Comparison of functional outcomes post-surgery and at 3, 6 and 12 months will enable assessment of recovery due to axonal regeneration.

Results shall assess the safety and feasibility of doing the study in emergency settings - enrolment and consent issues and assess effect size, this will provide sufficient information and, if successful, will lead to a definitive Randomised Control Trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Age >18.
* Cauda equina syndrome with bladder, bowel or sexual dysfunction (CES-I or CES-R) secondary to acute lumbar disc prolapse.
* Selected for emergency surgery.

Exclusion Criteria:

* No bladder, bowel or sexual dysfunction (Only bilateral radicular symptoms).
* Previous spinal surgery with risk of adhesions.
* Multilevel degeneration with inadequate safe space to pass epidural electrode.
* Pre-existent bladder, bowel or sexual dysfunction.
* History of peripheral neuropathy.
* Contraindications to neurostimulation (e.g. pacemaker, immune deficiency, uncontrolled diabetes, sepsis, active pressure sore, spinal cord stimulator in situ).
* Intraoperative CSF leak.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-09-08 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 6 months
  Recruitment rate of 50% or above will be considered sufficient for feasibility of conducting future RCT.
Pudendal Somatosensory Evoked Potentials (SEP) - amplitude (uV) | Post-operatively and at 3 months.
  In participants who do not recover autonomic function, Pudendal Nerve SEP will be performed to assess baseline conduction in residual neurons and recovery rate. Results at 3 months will be compared against baseline.
Pudendal Somatosensory Evoked Potentials (SEP) - latency (ms) | Post-operatively and at 3 months.
  In participants who do not recover autonomic function, Pudendal Nerve SEP will be performed to assess baseline conduction in residual neurons and recovery rate. Results at 3 months will be compared against baseline.
Stimulation parameters - Frequency (Hz) | At the time of the surgery and immediately post-op
  Intraoperative stimulation parameters will be set to the motor threshold - visually assessed motor response to stimulation. Post-operative stimulation parameters will be set according to patients response - sensation of motor contraction or paraesthesia. Default frequency is 20 Hz and can be modified in 10Hz increments. Descriptive analysis of these parameters shall enable optimisation of settings in future studies.
Stimulation parameters - Amplitude (mA) | At the time of the surgery and immediately post-op
  Intraoperative stimulation parameters will be set to the motor threshold - visually assessed motor response to stimulation. Post-operative stimulation parameters will be set according to patients response - sensation of motor contraction or paraesthesia. Amplitude is increased in 0.1mA increments until response is ascertained. Maximal safe amplitude is considered to be 15mA. Descriptive analysis of these parameters shall enable optimisation of settings in future studies.
Stimulation parameters - Pulse width (microseconds) | At the time of the surgery and immediately post-op
  Intraoperative stimulation parameters will be set to the motor threshold - visually assessed motor response to stimulation. Post-operative stimulation parameters will be set according to patients response - sensation of motor contraction or paraesthesia. Default pulse width is 100 microseconds and it can be adjusted in 10 microsecond increments. Descriptive analysis of these parameters shall enable optimisation of settings in future studies.

SECONDARY OUTCOMES:
Short Form Incontinence Questionnaire (SFIQ) | On admission and at 3, 6 and 12 months.
  The SFIQ consists of 5 items. Items 1 and 5 are Yes/No questions. Item 2 is an 8-question scale with answers ranging from 0 (best) to 3 (worst) each. Item 3 is a scale ranging from 1 (best) to 8 (worst). Item 4 is a scale ranging from 1 (best) to 6 (worst).
Arizona Sexual Experiences Scale (ASEX) | On admission and at 3, 6 and 12 months.
  The ASEX consists of 5 questions with answers from 1 (best) to 6 (worst)
Neurogenic Bowel Dysfunction (NBD) Questionnaire | On admission and at 3, 6 and 12 months.
  NBD is a 10-question item with a score range from 0 (best) to 47 (worst). A score of 0-6 is considered very minor, 7-9 minor, 10-13 moderate and 14+ severe.
Oswestry Disability Index (ODI) | On admission and at 3, 6 and 12 months.
  The ODI assesses disability related to back pain. It is a 10-question item, each scored from 0 (best) to 5 (worst). The total score is between 0 (best) and 50 (worst).
Rand SF-36 Questionnaire | On admission and at 3, 6 and 12 months.
  Rand Short Form Health Survey (SF-36) is a 36-question tool, developed at RAND as part of the Medical Outcomes Study. It assesses the quality of life in 9 categories (Physical functioning, Role limitations due to physical health, Role limitations due to emotional problems, Energy/fatigue, Emotional well-being, Social functioning, Pain, General health, Health change). Each category is scored from 0% (worst) to 100% (best).
Post-void bladder scan (PVBS) | At baseline, post-operative (x3) and at 3 months.
  PVBS assesses post-micturition bladder volume. Volume above 200mL suggests incomplete bladder emptying or retention. Trends in PVBS will be assessed post-operatively and at 3-month follow-up in patients with incomplete recovery following the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Marshall, PhD, Study Chair — University of Liverpool
Locations (1):
- The Walton Centre NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Majed AA, Neumann CM, Brushart TM, Gordon T. Brief electrical stimulation promotes the speed and accuracy of motor axonal regeneration. J Neurosci. 2000 Apr 1;20(7):2602-8. doi: 10.1523/JNEUROSCI.20-07-02602.2000. PMID 10729340
- [Background] Gordon T, Amirjani N, Edwards DC, Chan KM. Brief post-surgical electrical stimulation accelerates axon regeneration and muscle reinnervation without affecting the functional measures in carpal tunnel syndrome patients. Exp Neurol. 2010 May;223(1):192-202. doi: 10.1016/j.expneurol.2009.09.020. Epub 2009 Oct 1. PMID 19800329
- [Background] Juckett L, Saffari TM, Ormseth B, Senger JL, Moore AM. The Effect of Electrical Stimulation on Nerve Regeneration Following Peripheral Nerve Injury. Biomolecules. 2022 Dec 12;12(12):1856. doi: 10.3390/biom12121856. PMID 36551285
- [Background] Power HA, Morhart MJ, Olson JL, Chan KM. Postsurgical Electrical Stimulation Enhances Recovery Following Surgery for Severe Cubital Tunnel Syndrome: A Double-Blind Randomized Controlled Trial. Neurosurgery. 2020 Jun 1;86(6):769-777. doi: 10.1093/neuros/nyz322. PMID 31432080
- [Background] Wong JN, Olson JL, Morhart MJ, Chan KM. Electrical stimulation enhances sensory recovery: a randomized controlled trial. Ann Neurol. 2015 Jun;77(6):996-1006. doi: 10.1002/ana.24397. Epub 2015 May 4. PMID 25727139
- [Background] Barber B, Seikaly H, Ming Chan K, Beaudry R, Rychlik S, Olson J, Curran M, Dziegielewski P, Biron V, Harris J, McNeely M, O'Connell D. Intraoperative Brief Electrical Stimulation of the Spinal Accessory Nerve (BEST SPIN) for prevention of shoulder dysfunction after oncologic neck dissection: a double-blinded, randomized controlled trial. J Otolaryngol Head Neck Surg. 2018 Jan 23;47(1):7. doi: 10.1186/s40463-017-0244-9. PMID 29361981
- [Background] Rascon-Ramirez FJ. Spinal cord stimulation and cauda equina syndrome: Could it be a valid option? A report of two cases. Neurocirugia (Engl Ed). 2021 Feb 5:S1130-1473(21)00003-8. doi: 10.1016/j.neucir.2020.12.002. Online ahead of print. English, Spanish. PMID 33558146
- [Background] Sayanagi J, Acevedo-Cintron JA, Pan D, Schellhardt L, Hunter DA, Snyder-Warwick AK, Mackinnon SE, Wood MD. Brief Electrical Stimulation Accelerates Axon Regeneration and Promotes Recovery Following Nerve Transection and Repair in Mice. J Bone Joint Surg Am. 2021 Oct 20;103(20):e80. doi: 10.2106/JBJS.20.01965. PMID 34668879
- [Background] Woodfield J, Hoeritzauer I, Jamjoom AAB, Jung J, Lammy S, Pronin S, Hannan CJ, Watts A, Hughes L, Moon RDC, Darwish S, Roy H, Copley PC, Poon MTC, Thorpe P, Srikandarajah N, Grahovac G, Demetriades AK, Eames N, Sell PJ, Statham PFX; UCES Collaborators; British Neurosurgical Trainee Research Collaborative. Presentation, management, and outcomes of cauda equina syndrome up to one year after surgery, using clinician and participant reporting: A multi-centre prospective cohort study. Lancet Reg Health Eur. 2022 Nov 17;24:100545. doi: 10.1016/j.lanepe.2022.100545. eCollection 2023 Jan. PMID 36426378